CLINICAL TRIAL: NCT03974724
Title: Preterm Birth Prediction by Measurement of Biomarkers in Cervical Vaginal Fluid
Acronym: PBMBCVF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: ESCO Beijing Technologies Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: Preterm birth prediction
Record Dates: First submitted 2019-05-16; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Preterm Birth
Keywords: Preterm birth; Prediction; Cervical vaginal fluid
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collect cervical vaginal fluid in posterior fornix in pregnant women whose gestational age are 16 to 24 weeks that enrolled into this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the predictive value of 7 biomarkers cervical vaginal fluid on future preterm birth in pregnant women whose gestational age are 16 to 24 weeks.

DETAILED DESCRIPTION:
Preterm births (PTBs) refers to a delivery with a gestational age prior to 37 weeks, which can be divided into extreme PTBs (<28 weeks), early PTBs (28-32 weeks), and advanced PTBs (32-37 weeks). The prevalence of PTBs is on a global scale, with more than 1 million PTB per year in China (with a prevalence of 7%), ranking the second in the world. PTBs is the main cause of perinatal death. Meanwhile, premature infants are at higher risk of short-term or long-term complications such as respiratory distress syndrome and mental retardation, causing huge economic and mental burdens on families and society. Most PTBs are spontaneous or caused by premature rupture of membranes (PROM) while the precisely reason remains unknown. Effective early prediction of PTBs and timely intervention are key to reducing PTBs and improving adverse pregnancy outcomes. Current prediction methods for PTBs can be divided into the following three categories: risk factor assessment, cervical length measurement, and biomarkers. However, about half of premature pregnant women do not have high-risk factors, and only premature risk factors cannot accurately identify prematurely at-risk populations. Biomarkers such as fetal fibronectin (fFN) have a very high negative predictive value (more than 95%), but positive predictive value is low (with 200 ng/ml as a cut-off value, and fFN predicts a positive predictive value for preterm birth at <34 weeks gestation reaching only 37.7%). Other biomarkers such as hyperphosphorylated insulin-like growth factor binding protein-1 (phIGFBP1) and placenta α1 microglobulin (PAMG-1) were detected, but their predictive effects were still dissatisfactory.

Therefore, there is no currently effective screening method for predicting the occurrence of PTBs. How to accurately predict and diagnose PTBs is still an unsolved problem in obstetrics. Our previous study identified seven biomarkers in cervical vaginal fluid(CVF) that may be associated with preterm birth and preliminary validation in animal experiments, suggesting that biomarkers in selected CVF may be effective predictors of PTBs, but larger samples of clinical trials are required for validation.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18years
2. Between 16-24 weeks gestation
3. Signed informed consent

Note:The investigators also recruit pregnant women who have the following risk factors for preterm birth and meet the criteria for admission: uterine malformation, history of induction, history of premature birth, premature rupture of membranes, history of abortion, history of cervical conization and cervical cerclage, vaginal bleeding, cervical shortening, Multiple pregnancies - twins, triplets, polyhydramnios, smoking, drug use, placenta previa, pregnancy through assisted reproductive technology.

Exclusion Criteria:

1. Rupture of the membrane before sampling
2. Manual or ultrasound vaginal examination within 6 hours of sampling
3. Vaginal bleeding within 48 hours of sampling (significant vaginal bleeding)

Note: exclusion criteria for sample are listed as follow:

After the delivery results are verified, the samples are excluded according to the sample exclusion criteria and the samples that do not meet the criteria are excluded, including:

1. Therapeutic preterm birth
2. Samples of blood contamination
3. Progesterone treatment at the time of sampling
4. Situations that other researchers believe need to be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The investigators aim to recruit asymptomatic pregnant women visit their hospital whose gestational age are between 16 to 24 weeks.
Study Population: The investigators aim to recruit pregnant women visit their hospital whose gestational age are between 16 to 24 weeks and meet the criteria for inclusion during the study periods. The investigators introduce the study to those pregnant women who visit their hospital early after confirming pregancy till beyond the inclusion gestational age.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Preterm birth | At the time of delivery
  Preterm birth refers to delivery with the gestational age prior to 37 weeks

SECONDARY OUTCOMES:
Neonatal low birth weight(LBW) | At the time of delivery
  LBW is defined as birth weigh less than 2500g
respiratory distress syndrome(RDS) | At the time of delivery
  the number of neonatal RDS occurs in participants' newborns
neonatal ICU(NICU) admission | At the time of delivery
  the number of neonates admitted to NICU

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China